CLINICAL TRIAL: NCT02628665
Title: Two-arm Phase III Trial Comparing Different Time of Endoscopic Photodynamic Therapy on Esophageal and/or Gastric Cardiac Cancer
Brief Title: Clinical Study of Time Optimizing of Endoscopic Photodynamic Therapy on Esophageal and/or Gastric Cardiac Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Henan University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FirstHenanUST,cancer center
Record Dates: First submitted 2015-11-27; First posted 2015-12-11 (Estimated); Last update posted 2015-12-11 (Estimated); Status verified 2015-10

CONDITIONS: Stage I Esophageal Adenocarcinoma; Stage II Esophageal Adenocarcinoma; Stage III Esophageal Adenocarcinoma; Stage I Esophageal Squamous Cell Carcinoma; Stage II Esophageal Squamous Cell Carcinoma; Stage III Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Adenocarcinoma Of Esophagus; Esophageal Squamous Cell Carcinoma | interventions — Dihematoporphyrin Ether

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 24 to 48 hours group (Experimental): photosensitizer(photofrin): 2mg/kg, Diomed Surgical Diode Laser:400mv/cm irridiation 750 seconds, 24 to 48 hours: The injection of photosensitizer(photofrin) 24 to 48 hours light irradiation power.
  630 nm laser irradiation (DIOMED): The diseased tissue with laser irradiation in 1200 seconds.
  Interventions: Drug: photosensitizer(photofrin); Device: 630 nm laser irradiation (DIOMED)
- 48 to 72 hours group (Active Comparator): photosensitizer(photofrin): 2mg/kg, Diomed Surgical Diode Laser:400mv/cm irridiation 750 seconds, 48 to 72 hours: The injection of photosensitizer(photofrin) 48 to 72 hours light irradiation power.
  630 nm laser irradiation (DIOMED): The diseased tissue with laser irradiation in 1200 seconds.
  Interventions: Drug: photosensitizer(photofrin); Device: 630 nm laser irradiation (DIOMED)

INTERVENTIONS:
Drug: photosensitizer(photofrin) — photosensitizer(photofrin): 2mg/kg
  Other Names: photofrin
Device: 630 nm laser irradiation (DIOMED) — 630 nm laser irradiation (DIOMED): The diseased tissue with laser irradiation in 1200 seconds.
  Other Names: DIOMED

SUMMARY:
The therapy of photofrin PDT was effective in improving life quality of patients with advanced esophageal and/or gastric cardiac cancer and the time optimizing for employing laser irradiation was of great importance.The purpose of this study is to evaluate the clinical efficacy and adverse effects of Photodynamic Therapy (PDT) on esophageal and/or gastric cardiac cancer during different time after inject photofrin.

DETAILED DESCRIPTION:
The investigators plan to recruit the patients who were pathologically confirmed with esophageal squamous cell carcinoma or gastric cardia adenocarcinoma from the Oct.2015. The patients will be divided into two groups. Group 1: Following intravenous administration of photofrin at dose of 2 mg/kg.b.w. as the photosensitizer, 630 nm laser irradiation (DIOMED) with 400 mW/cm was applied on each part of tumor for 750 seconds through cylinder diffusing quartz fibers localizing in the biopsy channel of a flexible endoscope at 24th. Group 2: Following intravenous administration of photofrin at dose of 2 mg/kg.b.w. as the photosensitizer, 630 nm laser irradiation (DIOMED) with 400 mW/cm was applied on each part of tumor for 750 seconds through cylinder diffusing quartz fibers localizing in the biopsy channel of a flexible endoscope at 48th.

ELIGIBILITY:
Inclusion Criteria:

* In the esophagus, patients with severe dysplasia and carcinoma in situ
* The patients have not received the surgery or chemo-radiotherapy.
* Hb≥80g/L, absolute neutrophil count ≥1.5×109/L, Plt≥90×109/L, ALT、AST≤2.5*N,Cr≤1.5*N.
* Performance status score 0-2

Exclusion Criteria:

* pregnant, lactating women
* History of organ transplantation
* The peripheral nervous system disorders
* Severe infection
* Oral capecitabine who have difficulty with,such as dysphagia,The activities of digestive ulcer, Gastrointestinal bleeding
* Severe chronic diseases, such as, hepatopathy, nephropathy, respiratory disease,high blood pressure, diabetes.
* Other malignant tumor in recent 5 years.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-10; Primary Completion 2017-10 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Partial remission rate | 3 months
  Photodynamic therapy for 3 months after the review of gastroscope for pathologic examination, to check the response rate

SECONDARY OUTCOMES:
The recent incidence of adverse reactions | 7-10 days
  Observe 7-10 days postoperatively in patients with the ratio of pain and difficulty swallowing

CONTACTS AND LOCATIONS:
Overall Officials: Shegan Gao, Doctor, Study Chair — The First Affiliated Hospital of Henan University of Science and Technology; Tanyou Shan, Master, Study Director — The First Affiliated Hospital of Henan University of Science and Technology; Caihong Dong, Master, Principal Investigator — The First Affiliated Hospital of Henan University of Science and Technology; Xiaozhi Yuan, Master, Principal Investigator — The First Affiliated Hospital of Henan University of Science and Technology; Lin Guo, Bachelor, Principal Investigator — The First Affiliated Hospital of Henan University of Science and Technology; Lijuan Zhang, Bachelor, Principal Investigator — The First Affiliated Hospital of Henan University of Science and Technology; Gailin Wang, Bachelor, Principal Investigator — The First Affiliated Hospital of Henan University of Science and Technology
Locations (1):
- The First Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan, China

REFERENCES:
- [Background] Lindenmann J, Matzi V, Neuboeck N, Anegg U, Baumgartner E, Maier A, Smolle J, Smolle-Juettner FM. Individualized, multimodal palliative treatment of inoperable esophageal cancer: clinical impact of photodynamic therapy resulting in prolonged survival. Lasers Surg Med. 2012 Mar;44(3):189-98. doi: 10.1002/lsm.22006. Epub 2012 Feb 14. PMID 22334351
- [Background] Yano T, Muto M, Minashi K, Iwasaki J, Kojima T, Fuse N, Doi T, Kaneko K, Ohtsu A. Photodynamic therapy as salvage treatment for local failure after chemoradiotherapy in patients with esophageal squamous cell carcinoma: a phase II study. Int J Cancer. 2012 Sep 1;131(5):1228-34. doi: 10.1002/ijc.27320. Epub 2012 Mar 2. PMID 22024814